CLINICAL TRIAL: NCT05888597
Title: Effect of L-menthol on Breathlessness and Exercise Capacity in Chronic Obstructive Pulmonary Disease: a Randomized
Brief Title: Efficacy of L-menthol on Breathlessness in Chronic Obstructive Pulmonary Disease
Acronym: Ment-COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Ment-COPD
Record Dates: First submitted 2023-05-02; First posted 2023-06-05 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Menthol

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized (ratio 1:1), double-blinded, placebo-controlled, crossover trial (RCT) design
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol (Experimental): In the trial, 30 minutes prior to performing submaximal CPET, participants will be administered, L-menthol patch which will be attached to the inside of a facemask that is connected to the breathing circuit.
  Interventions: Drug: L-menthol
- Placebo (Placebo Comparator): For placebo, the patch will contain a similarly patch with strawberry scent.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-menthol — (Sigma-Aldrich, St. Louis, US)
  Arms: Menthol
Other: Placebo — Strawberry scent (Sigma-Aldrich, St. Louis, US)
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of L-menthol on breathlessness in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Breathelssness (Dyspnea) is a cardinal symptom in patients with chronic obstructive pulmonary disease (COPD), often triggered by daily-life physical activities. Despite optimal treatment of the underlying disease, many patients still suffer from chronic and disabling dyspnea for many years, leading to exercise intolerance, and worse morbidity and mortality. To date, an effective pharmacologic treatment to relieve chronic dyspnea is lacking. Recent pilot data support that inhaled L-menthol can markedly decrease laboratory-induced dyspnea in COPD patients, likely through increased afferent feedback of airflow in the airways by inducing a cooling sensation through olfactory stimulation. The aim of this study is therefore to assess the effectiveness and mechanisms of inhaled menthol for relief of chronic dyspnea in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written consent to participate in the study
* Diagnosis of COPD confirmed by spirometry and a FEV1 < 80% of predicted post bronchodilator at baseline
* age 18 years or older
* able to cycle
* able to understand and talk Swedish to participate in the study procedures, as judged by the Investigator.

Exclusion Criteria:

* Resting peripheral oxygen saturation (SpO2) < 92%
* hospitalization or clinical instability during the last four weeks
* treatment with supplementary oxygen at rest or during exercise
* contraindication to exercise testing in accordance with clinical practice guidelines
* expected survival shorter than six months as judged by the Investigator
* medical conditions including congestive heart failure, acute coronary artery disease, neuromuscular diseases, severe psychiatric illness, and olfaction disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Breathlessness intensity | Through study completion, up to 1 year
  The difference between treatment conditions in dyspnea intensity (Borg CR10 scale) at iso-time.

SECONDARY OUTCOMES:
Dyspnea unpleasantness | Through study completion, up to 1 year
  The difference between treatment conditions in dyspnea unpleasantness (Borg CR10 scale) at iso-time.
Total time | Through study completion, up to 1 year
  Time to the limit of tolerance (s) (tLIM)
Exercise capacity | Through study completion, up to 1 year
  V'O2 (aerobic exercise capacity, absolute and in %pred)
Work load | Through study completion, up to 1 year
  Workload (W and %pred)
Minute ventilation | Through study completion, up to 1 year
  Minute ventilation
Tidal volume (VT) | Through study completion, up to 1 year
  Tidal volume (VT)
Ventilatory reserve | Through study completion, up to 1 year
  Ventilatory reserve, defined as maximal voluntary ventilation (MVV) - VE
Cardiac reserve | Through study completion, up to 1 year
  Cardiac reserve, evaluated using the predicted peak heart rate
Inspiratory capacity | Through study completion, up to 1 year
  Inspiratory capacity (IC) during exercise
Breathing frequency | Through study completion, up to 1 year
  Breathing frequency during exercise
Peak dyspnea intensity | Through study completion, up to 1 year
  Dyspnea intensity at peak exercise (Borg CR10)
Leg discomfort | Through study completion, up to 1 year
  Leg discomfort (Borg CR10)
Anaerobic threshold | Through study completion, up to 1 year
  Timing (and V'O2) of the anaerobic threshold (AT)
Ventilatory efficacy | Through study completion, up to 1 year
  Efficacy of ventilation (VE/V'CO2-slope)
Respiratory exchange ratio | Through study completion, up to 1 year
  Respiratory exchange ratio (RER), defined as V'CO2/V'O2
Saturation | Through study completion, up to 1 year
  O2-saturation
Stop reason | Through study completion, up to 1 year
  Causes of stopping the test
Adverse events | Through study completion, up to 1 year
  Any adverse events during the test

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Ahmadi, MD, PhD, Principal Investigator — Region Skåne
Locations (1):
- Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT05888597/SAP_000.pdf